CLINICAL TRIAL: NCT02675608
Title: Vaccine Efficacy in Diabetic and Elderly Patients
Status: Completed | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Louisiana Clinical and Translational Science Center (Other)
Responsible Party: Principal Investigator, Elizabeth Norton, Assistant Professor, Tulane University
Other Study IDs: 15-727936
Record Dates: First submitted 2016-01-22; First posted 2016-02-05 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Inflammation
Keywords: vaccine efficacy; inflammation; aging; Type 2 Diabetes Mellitus; flu vaccine
MeSH Terms: conditions — Inflammation; Diabetes Mellitus, Type 2; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — plasma, serum, PBMCs, urine, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Year 1 Group 1: They are between 18-65 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; have no history of immunodeficiency or weakened immunologic function; do not have diabetes; and do not have chronic HIV or hepatitis B or C infection.
  Interventions: Biological: Influenza Virus Vaccine
- Year 1 Group 2: They are ≥65 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; have no history of immunodeficiency or weakened immunologic function; do not have diabetes; and do not have chronic HIV or hepatitis B or C infection.
  Interventions: Biological: Influenza Virus Vaccine
- Year 1 Group 3: They are between 18-65 years of age, are currently diabetic, and meet the criteria listed above for not diabetic subjects in Group 1, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).
  Interventions: Biological: Influenza Virus Vaccine
- Year 1 Group 4: They are ≥65 years of age, are currently diabetic, and meet the criteria listed above for non-diabetic subjects in Group 2, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).
  Interventions: Biological: Influenza Virus Vaccine
- Year 1 Group 5: They are between 35-50 years of age, meet the criteria listed above for non-diabetic subjects in Group 1, with the exception of chronic HIV with or without hepatitis B or C infection, and have current medical history of CD4 T-cell counts 300-800.
  Interventions: Biological: Influenza Virus Vaccine
- Year 2 Group 1: They are between 18-64 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; do not have diabetes.
- Year 2 Group 2: They are ≥65 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; do not have diabetes.
- Year 2 Group 3: If they are between 18-64 years of age, are currently diabetic, and meet the criteria listed above for not diabetic subjects in Group 1, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).
- Year 2 Group 4: If they are ≥65 years of age, are currently diabetic, and meet the criteria listed above for non-diabetic subjects in Group 2, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).

INTERVENTIONS:
Biological: Influenza Virus Vaccine — On the first visit, subjects are vaccinated with the 2015-2016 seasonal flu vaccine.
  Other Names: FLUVIRIN® NDC 66521-118-11
  Groups: Year 1 Group 1; Year 1 Group 2; Year 1 Group 3; Year 1 Group 4; Year 1 Group 5

SUMMARY:
This study evaluates the effectiveness of the seasonal flu vaccine in adults of different ages and diabetic disease statuses. These studies will help our understanding of how chronic inflammatory diseases impact immunologic function and future research on mitigation strategies.

DETAILED DESCRIPTION:
Our goal is to determine if an individual's level of inflammation determines their response to vaccination. The aging process and certain diseases, like type-2 diabetes, have been characterized as chronic inflammatory conditions. These individuals have higher rates of influenza disease and health care costs; hence, yearly vaccination is recommended. There is a paucity of information comparing vaccination in these high-risk groups and identifying biomarkers that can predict vaccine efficacy. The investigators hypothesize that elderly and diabetic patients have reduced responses to seasonal influenza vaccination that are inversely proportional to their level of chronic inflammation. In this pilot proposal, the investigators will examine adult and elderly diabetic and non-diabetic adults for markers of inflammation and vaccine efficacy before and after influenza vaccination. These studies will help our understanding of how chronic inflammatory diseases impact immunologic function and future research on mitigation strategies.

ELIGIBILITY:
Year 1 Inclusion Criteria:

* Group 1: Must be 18-64 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; have no history of immunodeficiency or weakened immunologic function; do not have diabetes; and do not have chronic HIV or hepatitis B or C infection.
* Group 2: Must be ≥65 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; have no history of immunodeficiency or weakened immunologic function; do not have diabetes; and do not have chronic HIV or hepatitis B or C infection.
* Group 3: Must be between 18-64 years of age, are currently diabetic, and meet the criteria listed above for not diabetic subjects in Group 1, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).
* Group 4: Must be ≥65 years of age, are currently diabetic, and meet the criteria listed above for non-diabetic subjects in Group 2, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).
* Group 5: Must be between 35-50 years of age, meet the criteria listed above for non-diabetic subjects in Group 1, with the exception of chronic HIV with or without hepatitis B or C infection, and have current medical history of CD4 T-cell counts 300-800.

Year 1 Exclusion Criteria:

* a history of sensitivity to any of the vaccine components or to influenza vaccine
* a history of Guillain-Barré syndrome
* a history of known or suspected impairment of immunologic function outside of criteria described in the inclusion criteria, including clinically significant liver disease, arthritis, moderate to severe renal (kidney) disease, and ongoing infections
* a history of a bleeding disorder or received anticoagulants within the last 3 weeks
* received the influenza vaccine in the past 6 months or any other vaccines within the last 3 months
* received immunosuppressive therapy within the last 6 months
* received long-term systemic corticosteroid therapy for more than 2 consecutive weeks within 3 months
* received blood or blood-derived products within the last 3 months
* a daily aspirin intake of >81mg
* a blood pressure >150/95 at screening

Year 2 Inclusion Criteria:

Group 1: They are between 18-64 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; do not have diabetes.

Group 2: They are ≥65 years of age, are medically stable and ambulatory; have no active systemic or serious concurrent illness; do not have diabetes.

Group 3: If they are between 18-64 years of age, are currently diabetic, and meet the criteria listed above for not diabetic subjects in Group 1, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).

NOTE: Current diabetes is defined by patient report of physician diagnosis. Subjects with a history of diabetes which has resolved and no longer requires therapy are not considered to have current diabetes, e.g, women with a history of gestational diabetes, steroid-induced or medication-induced.

Group 4: If they are ≥65 years of age, are currently diabetic, and meet the criteria listed above for non-diabetic subjects in Group 2, with the exception of having pre-diagnosed type-2 diabetes mellitus (e.g., a history of hemoglobin A1C or HbA1C scores of > 6.5%).

Year 2 Subjects will be excluded if they have any of the following:

* a history of known or suspected impairment of immunologic function, including clinically significant liver disease, arthritis, moderate to severe renal (kidney) disease, HIV, and ongoing infections
* a history of a bleeding disorder or received anticoagulants within the last 3 weeks
* a history of heart failure
* a history of receiving immunosuppressive therapy within the last 6 months
* a history of receiving long-term systemic corticosteroid therapy for more than 2 consecutive weeks within 3 months
* a history of receiving blood or blood-derived products within the last 3 months
* a daily aspirin intake of >325mg
* are pregnant

There are no inclusion/exclusion criteria based on race. Each group will have a targeted enrollment of 50% female to male ratio. Women cannot be pregnant or breastfeeding. There will be no children involved in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In Year 1 during the 2015-16 flu season, subjects were recruited from the New Orleans metropolitan area through flyers, radio ads, internet ads, social media, and doctor referrals and vaccinated. These subjects were administered the 2015-16 flu vaccine as part of their study visit. In Year 2 during the 2016-17 flu season, subjects were recruited from populations immediately prior or following receiving the flu vaccine at vaccination events, including senior living facilities contracted with the CTU and Tulane University vaccination events for faculty, staff, students.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in HAI titer from day 0 to day 30 (+/- 4 days) | 30 days (+/- 4 days)
  Blood samples collected days 0 and 30 will be evaluated and compared for flu antibodies using the standards HAI assay with individual virus strains contained in vaccine.

SECONDARY OUTCOMES:
Inflammatory Soluble Factor and Cellular Analysis | day 0
  Inflammatory Analysis will be performed on day 0 samples. Soluble factors in the serum will be analyzed using flow cytometry and bioplex. This analysis will evaluate cellular proliferation, senescence, and recognized inflammatory subsets within myeloid and lymphoid cell subsets.
Inflammatory Soluble Factor and Cellular Analysis additional measurements | day 30 (+/- 4 days)
  Additional Inflammatory Analysis will be performed on day 30 samples. Soluble factors in the serum will be analyzed using flow cytometry and bioplex. This analysis will evaluate cellular proliferation, senescence, and recognized inflammatory subsets within myeloid and lymphoid cell subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Norton, MPH, PhD, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane Clinical Translational Unit, New Orleans, Louisiana, United States